CLINICAL TRIAL: NCT03723629
Title: Progression of Untreated Pulmonary Ground Glass Opacity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2018-137R
Record Dates: First submitted 2018-10-20; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
Keywords: Ground glass opacity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pulmonary GGO: Patients with pulmonary GGO.
  Interventions: Other: No intercention

INTERVENTIONS:
Other: No intercention — No intercention

SUMMARY:
In this study, about 2000 GGO patients will be included for a 5-year follow-up. The aim of this study is to elucidate the biological nature of pulmonary GGO lesion and provide evidence for GGO treatment.

ELIGIBILITY:
Inclusion Criteria:

* 35-80 years' old
* found pulmonary GGO with chest CT scan and CT follow-up after 3 months shows that the GGO remains
* Diameter of GGO > 5mm and < 3cm
* Solid component of GGO in pulmonary window < 5mm
* signed informed consent form

Exclusion Criteria:

* receiving immunosuppressor or steriods
* receiving chemo- or radio- therapy
* can not receive regular follow-up

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic out patients of thoracic surgery.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline GGO diameter | 6 months, 1year, 2 years, 3 years, 4 years and 5 years
  Changes from baseline GGO diameter
Changes from baseline GGO CT index. | 6 months, 1year, 2 years, 3 years, 4 years and 5 years
  Changes from baseline GGO CT index.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided